CLINICAL TRIAL: NCT00163761
Title: A Multicentre Phase II Study of Risk-adjusted Outpatient-based Salvage Therapy for Patients With Relapsed and Refractory Lymphoma
Brief Title: Efficacy Study of Outpatient Therapy for Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AH226/02
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Disease
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma | interventions — Gemcitabine; Vinorelbine; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Commence VGF treatment (Active Comparator): Drug. Vinorelbine, gemcitabine and filgrastim 21 day cycle
  Interventions: Drug: gemcitabine, vinorelbine, filgastrim
- Commence F-GIV treatment (Active Comparator): Drug. Gemcitabine, ifosfamide, Vinorelbine and filgrastim 21 day cycle
  Interventions: Drug: gemcitabine, vinorelbine, ifosfamide, filgastrim

INTERVENTIONS:
Drug: gemcitabine, vinorelbine, ifosfamide, filgastrim — Drug
  Arms: Commence F-GIV treatment
Drug: gemcitabine, vinorelbine, filgastrim — Drug
  Arms: Commence VGF treatment

SUMMARY:
This is a Phase II trial evaluating the efficacy (overall response rate) of a risk-adjusted outpatient based approach to lymphoma salvage therapy with vinorelbine, gemcitabine and pegfilgrastim and/or gemcitabine, ifosfamide, vinorelbine and pegfilgrastim.

DETAILED DESCRIPTION:
Lymphoma has been increasing in incidence annually for the past several decades and the majority of patients relapse after first line therapy. A variety of 'salvage chemotherapy' treatments are available that are usually inpatient-based treatments associated with significant haematological toxicity. Furthermore, all patients are treated in the same manner despite the fact that some patients will do well irrespective of the type of salvage therapy whereas others will do badly no matter what is done. During 2001-2002 we undertook a pilot study in 40 such patients using an outpatient-based salvage therapy with 2 newer chemotherapy drugs, vinorelbine and gemcitabine. Over 75% of all treatments were successfully delivered on an outpatient basis with response rates similar to historical controls. We now propose to expand on these initial findings by modifying the outpatient approach for those patients with less favourable prognostic features, that is, patients will be stratified to differing therapies but with the majority still receiving the proven vinorelbine-gemcitabine combination.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* relapsed or primary refractory non-Hodgkin's lymphoma (NHL) or Hodgkin's Disease (HD)
* ECOG 0 - 2
* written informed consent

Exclusion criteria:

* Intention to proceed with any form of transplant therapy following fewer than 2 cycles of protocol salvage therapy
* bilirubin > 50μmol/litre unless secondary to lymphoma
* creatinine > 2 x upper limit of normal unless secondary to lymphoma, absolute neutrophil count <0.5 x 109/litre and / or platelets < 50 x 109/litre unless secondary to lymphoma
* relapse within 6 months of a prior transplant procedure (autologous or allogeneic)
* known sensitivity to E coli derived preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy (overall response rate) of a risk-adjusted outpatient-based approach to lymphoma salvage therapy with VGF (vinorelbine, gemcitabine and pegfilgrastim) and/or F-GIV (gemcitabine, Ifosfamide, vinorelbine and pegfilgrastim). | After two cycles and after four cycles

SECONDARY OUTCOMES:
To evaluate safety, | Days 1 and 8 for every cycle, days 10,12,14, and 16 for first cycle.
relapse free survival, | After 2 cycles, 4 cyles and every 3 or 4 months for 12 months. Then every 6 months until disease progression
overall survival, | every 3 or 4 months for 12 months. Then every 6 months.
and planned dose-on-time. | After two cycles and after four cycles

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spencer, Assoc. Prof, Study Chair
Locations (10):
- Australia (10):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal North Shore Hospital, Sydney, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Frankston Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Fremantle Hospital, Fremantle, Western Australia